CLINICAL TRIAL: NCT04863911
Title: Comparative Study Between CT Arthrography and MRI Arthrography in Detection of Intra-articular Hip Pathology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nafisa Desouky Mohamed Hussein, specialist of radiology Assuit University Hospitals, Assiut University
Other Study IDs: CTA vs MRA in hip pathology
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Hip Disease
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: combined CT and MRI — 1 mL of gadolinium-diethylenetriamine pentaacetic acid (Gd-DTPA) will be diluted with 100 mL of saline; 8 mL of this will be mixed with 7 mL of iodine solution (340 mg/cc) and 3 mL of lidocaine 2% and injected under ultrasonographic guidance.
  The fixed US-guided technique, the needle will be inserted into the needle guide hole and directed toward the hip joint, targeting the femoral head-neck junction. The volume injected varies from 10 to 20 mL, with a mean of 15 mL.
  Ideally CT should be performed immediately after the injection and MR should be performed within 90 minutes after the initial injection.

SUMMARY:
The aim of this work is to compare the role of CT hip arthrography to MR arthrography in the detection of intra-articular hip pathology.

DETAILED DESCRIPTION:
The hip joint is a ball-and-socket synovial joint designed to allow multi-axial motion while transferring loads between the upper and lower body. The acetabular rim is lined by fibrocartilage (labrum), which adds depth and stability to the femoro-acetabular joint. The articular surfaces are covered by hyaline cartilage that dissipates shear and compressive forces during load bearing and hip motion.

Various anatomical factors make the investigation of suspected intra-articular hip pathology challenging. Lesions of the labrum, cartilaginous lesions, femoro-acetabular impingement (FAI), and intra-articular foreign bodies are the most common intra-articular pathology , others causes of intra-articular hip pain include ligamentum teres rupture, degenerative changes, arthritis (inflammatory, infectious, etc.), and synovial proliferative disorders.

The labrum is a fibrocartilaginous triangular-shaped incomplete ring that surrounds the bony acetabulum. The labrum increases the depth of the acetabulum, thereby assisting hip stability and distributing hip load. It also seals the hip joint, helping to maintain synovial fluid within the central compartment and becoming a mechanical stabilizer. The articular cartilage of the acetabulum has a horseshoe shaped appearance with an opening at the acetabular notch, is not as thick as in other joints such as the knee. Hip cartilage in adults has been estimated to be between 1 and 2 mm in thickness. Thus, plain MRI and CT have limited value in assessing labral and articular cartilage disorders. Acetabular labral tears are a potential source of hip pain in young adults. Many underlying conditions may predispose to labral degeneration and tear including prior trauma, femoroacetabular impingement (FAI), developmental dysplasia of the hip (DDH), capsular laxity, and congenital abnormalities involving the axis of the joint such as acetabular retroversion and anteversion. Labral tears rarely occur in the absence of bony abnormalities and that neglecting these underlying structural abnormalities may result in treatment failure. FAI is defined as an abnormal contact between the femoral head and the acetabulum that limits normal range of motion. Although two types were defined (pincer when focal or general acetabular over coverage occurs and cam when there is an abnormal contact between the femoral head-neck junction and the anterior acetabulum), most patients have mixed types.

Arthroscopy is the gold standard for clarifying diagnostic dilemmas but is an invasive procedure with possible complications and cannot be applied to every patient with suspected but not established hip pathology. Thus, imaging may play an important role in planning joint-preserving treatment options in those cases and thus preventing early hip osteoarthritis.

The diagnosis of a labral tear is made on CT arthrography (CTa) and MR arthrography (MRa) when contrast fluid gets inside the labrum. Fluid-sensitive sequences are needed on MRa to detect intrasubstance labrum changes, especially those that do not extend to the articular surface. Unless calcified, these changes are missed on CTa.

Much of the radiology literature has focused on the use of MRa of the hip to detect labral and cartilage pathology. Both non-contrast MRI and MRa have limitations in terms of spatial resolution, which can make the detection of subtle labral and cartilage pathology challenging.

CT arthrography (CTa) with its superior spatial resolution offers several advantages over plain MRI for the evaluation of articular cartilage. Image acquisition at a submillimeter scale together with the availability of multiplanar reformations can reveal early intraarticular changes that are poorly detected on plain MRI. Although Multidetector Computed Tomography (MDCT) has higher spatial resolution than MR, it has significantly lower contrast resolution, and thus labra and extraarticular pathology are not evaluated to the same extent.

CTa may be indicated in cases of MR incompatibility and MR contraindications. So in our study we try prospectively to evaluate the diagnostic value of CTa in comparison to MRa in detection of intraarticular hip pathology

ELIGIBILITY:
Inclusion Criteria:

* 60 consecutive patients presenting with clinical and routine imaging suggestive of intraarticular hip pathology.
* patients must be accept the intraarticular hip injection of contrast.

Exclusion Criteria:

* Any general contraindication of MRI in some cases as presence of anti-paramagnetic substance as pacemakers aneurysm clips, metallic cochlear implants
* Severely ill patients or those with claustrophobia
* Any general contraindications to radiation in some cases such as pregnancy at first trimester.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of different sex and age groups presenting to the Radiology department with clinical and routine imaging suggestive of intraarticular hip pathology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 week
  Sensitivity refers to true positive rate, the percentage of patients with actual illness who was correctly diagnosed in overall patients by each of CT arthrography and MRI arthrography. High sensitivity indicated high correct rate in diagnosis of intra-articular hip pathology.

SECONDARY OUTCOMES:
Specificity | 1 week
  Specificity refers to true negative rate, the percentage of patients with actual disease-free who are correctly judged as disease-free according to the diagnostic criteria. The high specificity indicates high accuracy of diagnosis.
positive predictive value | 1 week
  Positive predictive value refers to the proportion of patients with actual illness among all positive cases, can reflect the possibility of affecting target disease in patients with positive screening test result.
Negative predictive value | 1 week
  Negative predictive value refers to the proportion of patients with negative screening test result who do not suffer from diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Mohammad, A. Professor, Study Director — Diagnostic radiology department Assiut university hospital; Noha Attia, Lecturer, Study Director — Diagnostic radiology department Assiut university hospital

REFERENCES:
- [Result] Llopis E, Fernandez E, Cerezal L. MR and CT arthrography of the hip. Semin Musculoskelet Radiol. 2012 Feb;16(1):42-56. doi: 10.1055/s-0032-1304300. Epub 2012 Mar 23. PMID 22447236
- [Result] Perdikakis E, Karachalios T, Katonis P, Karantanas A. Comparison of MR-arthrography and MDCT-arthrography for detection of labral and articular cartilage hip pathology. Skeletal Radiol. 2011 Nov;40(11):1441-7. doi: 10.1007/s00256-011-1111-9. Epub 2011 Feb 6. PMID 21298428
- [Result] Schneider G, Massmann A, Fries P, Kusma M, Dienst M. [Magnetic resonance tomography and arthrography of the hip joint]. Orthopade. 2006 Jan;35(1):22-6, 28-32. doi: 10.1007/s00132-005-0890-x. German. PMID 16322973